CLINICAL TRIAL: NCT06694168
Title: Efficacy of the Entire Papilla Preservation Technique With and Without the Use of L-PRF as a Regenerative Material for the Treatment of Infrabony Defects: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of the Entire Papilla Preservation Technique With and Without the Use of L-PRF as a Regenerative Material for the Treatment of Infrabony Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEC2024045
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: Periodontal Regeneration; Minimally Invasive Surgical Technique; Platelet Rich Fibrin; Microsurgery; Periodontal Intrabony Defect; Periodontal Disease
Keywords: Periodontitis; Guided Tissue Regeneration; Microsurgery; Bone Regeneration; Treatment Outcome; Intrabony defect; minimally invasive surgical technique; Entire papilla preservation
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: To calculate the sample size, statistically significant EVA values were taken from a previous series of cases in the same line of research. The values were analyzed using STATA software, resulting in an N of 26 patients (26 defects). Finally, a final N of 30 defects to be treated was established (1 defect per patient), overestimating the initial N in case of possible losses during the follow-up period. If there is more than one site per patient that needs to be treated, it will be decided randomly which site will be included in the study, treating all sites with the same technique.
  The sample was randomized using the digital STATA software, separating the sample into sites to be treated using the EPP technique with defect filling using LPRF (15 defects) and sites to be treated with the same technique but without LPRF (15 defects).
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPP with L-PRF as a filling material (Experimental): This group will have the infrabony defect treated with the use of an EPP minimally invasive technique and the defect will be filled with L-PRF.
  Interventions: Procedure: Periodontal Regeneration, clinical and radiographic results, modified minimal invasive surgery; Procedure: REGEND001 Autologous Therapy Product
- EPP with no defect filling material (Active Comparator): This group will have the infrabony defect treated with the use of an EPP minimally invasive technique, but the defect will not be filled with L-PRF.
  Interventions: Procedure: Periodontal Regeneration, clinical and radiographic results, modified minimal invasive surgery

INTERVENTIONS:
Procedure: Periodontal Regeneration, clinical and radiographic results, modified minimal invasive surgery — The Entire Papilla Preservation Technique (EPP) is a minimally invasive surgical approach for the treatment of intraosseous defects allowing access to the defect maintaining the integrity of the interproximal papilla. Studies have evaluated its efficacy for the regeneration of intraosseous periodontal defects with or without the use of regenerative biomaterials to fill the defect.
Procedure: REGEND001 Autologous Therapy Product — L-PRF is an autologous concentrate of platelet- and leukocyte-rich fibrin derived from blood, which through a centrifugation process allows to stimulate, improve and accelerate healing. The growth factors in the concentrates, together with pro-inflammatory and anti-inflammatory molecules, actively participate in the stimulation of the processes associated with tissue and bone repair and regeneration. Due to its high content of fibrin, platelets, leukocytes, monocytes and stem cells, L-PRF acts in immune regulation by controlling inflammation, with a continuous release of growth factors and presents an analgesic effect, which gives greater postoperative comfort to the patient. In addition, being an autologous product, it greatly reduces the risk of infection or rejection by the patient. Due to its beneficial biological effects, low costs and ease of preparation its use as a filling material in intraosseous defects will be evaluated.
  Arms: EPP with L-PRF as a filling material

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of using L-PRF (leukocyte and platelet rich fibrin clot) as an autologous filling material in conjunction with the EPP (entire papilla preservation) technique for the treatment of interproximal intraosseous periodontal defects, compared to the same technique without L-PRF regarding clinical periodontal parameters and obtained radiographic parameters. It will also report possible postoperative complications and evaluate postoperative sensitivity. The main questions it aims to answer is:

• What is the effectiveness of LPR-F in conjunction with a complete papilla preservation (EPP) technique for the treatment of intrabony periodontal defects in CESA (health care center) patients in terms of clinical and radiographic periodontal parameters compared to the use of the same technique without L-PRF?

A non-randomized controlled clinical trial will be conducted on patients at CESA of the Universidad de los Andes. In 30 patients, 30 periodontal defects associated with a pocket with probing depths equal to or greater than 6 mm will be treated using the complete papilla preservation technique, either with L-PRF filling or without any filling material, assigned randomly to each intervention (15 participants in each group). Researchers will evaluate clinical and radiographic parameters at baseline and 6 months post-surgery. Patients will report their level of pain 24 hours and 7 days after surgery.

DETAILED DESCRIPTION:
Periodontitis is an infectious disease of bacterial origin that leads to a slow and progressive loss of periodontal attachment, resulting in the destruction of supporting tissues and the formation of periodontal pockets. These pockets can be classified as suprabony or intrabony, with the latter being those where the bottom of the pocket is apical to the level of the adjacent alveolar bone and the bone loss presents a vertical pattern. Intraosseous defects affect 36% of periodontal patients and are particularly challenging to treat due to their association with greater loss of periodontal support, increased clinical attachment loss, deeper probing depths, greater tooth mobility, and functional consequences for the patient; thus, they have a less favorable prognosis and response to non-surgical periodontal treatment.

Lang et al. established that periodontal defects can be successfully treated with non-surgical therapy, limiting additional surgical interventions to sites with an initial probing depth of 6 mm or more, or to advanced periodontal lesions that, after a successful etiological phase, still retain residual pockets ≥ 6 mm. Given this, surgical periodontal therapy becomes a therapeutic alternative for intraosseous defects associated with advanced periodontal destruction, aiming to reduce tooth loss over time, recover lost periodontal support, and improve patient's quality of life.

Different surgical alternatives have been developed to enhance short- and long-term clinical outcomes in teeth with infrabony defects and reduced periodontal support. If the contour of the existing bone and the number of remaining bony walls are favorable, regenerative surgical therapy could successfully regenerate bone up to the level of the alveolar crest. The use of materials such as a demineralized allogeneic bone matrix in guided tissue regeneration has shown to achieve reductions in probing depths, gains in clinical attachment level, and filling of treated defects compared to defect instrumentation through open flap debridement.

However, these treatment modalities are sensitive to technique, and their outcomes depend on various factors including patient-dependent factors such as plaque control and smoking habits; site-specific factors, such as defect morphology; and factors inherent to the surgical techniques employed. Consequently, the failure of conventional surgical techniques, such as early exposure of the regenerated area, has been reported in the scientific literature and is even more frequent with the use of membranes and bone substitutes.

In light of this, innovations in flap design and soft tissue management have reduced failures associated with early wound closure. Surgical techniques such as simplified papilla flap and modified techniques, minimally invasive surgical technique (MIST), and modified minimally invasive surgical technique (M-MIST) have been designed to protect the regeneration site and facilitate the stability of the blood clot.

Recently, the complete papilla preservation technique has been proposed for treating intraosseous defects through regeneration, with a surgical approach designed to fully preserve the integrity of the interdental papilla, thus achieving an optimal environment for wound healing. Full access to the defect is achieved through a tunnel incision with vertical release and the elevation of a short flap on the contralateral side of the tooth associated with the defect. Then, enamel matrix derivatives and bone substitutes are applied to the defect to promote periodontal regeneration at the site. Although the evidence supporting the success of this technique is limited, in 2020 Aslan et al. compared the outcomes of using this technique with and without biomaterials for filling the defect. They reported no statistically significant differences in clinical attachment gain, probing depth reduction, or increase in gingival recession between the groups treated with the complete preservation technique and filling material or with the technique alone, respectively. They concluded that the use of this technique with and without regeneration materials resulted in improvements in the clinical and radiographic parameters of the treated defects.

The search for different materials with regenerative potential has led to the use of L-PRF (leukocyte and platelet rich fibrin), an autologous platelet-rich fibrin and leukocyte concentrate derived from blood that stimulates, enhances, and accelerates healing through a centrifugation process. The growth factors present in the concentrates, along with pro-inflammatory and anti-inflammatory molecules, actively participate in the stimulation of processes associated with tissue and bone repair and regeneration. Due to its high content of fibrin, platelets, leukocytes, monocytes, and stem cells, L-PRF regulates the immune response by controlling inflammation, with a continuous release of growth factors and an analgesic effect, providing greater postoperative comfort to the patient. Additionally, being an autologous product significantly reduces the risk of infection or rejection by the patient. Due to its beneficial biological effects, low costs, and ease of preparation, it is widely used in the periodontal surgical field.

One of the goals of treating infrabony defects is the regeneration of soft and hard tissues, which is why using a complete papilla preservation surgical technique along with L-PRF as a biomaterial is a minimally invasive alternative to achieve this. The properties of L-PRF mentioned above will improve the biological conditions of the site and reduce postoperative complications, making its use in regenerative periodontal therapy worthy of deeper investigation. This is even more relevant given the lack of studies reporting the use of L-PRF associated with this surgical technique.

The aim of this study is to evaluate the efficacy of using a papilla preservation technique for the treatment of interproximal infrabony periodontal defects, with and without the additional use of L-PRF, concerning clinical and radiographic parameters. Its importance is based on the need in the field of periodontology to find minimally invasive, effective, and low-cost surgical techniques with the least amount of postoperative complications that allow for the treatment of infrabony defects in teeth affected by severe periodontitis, a growing public health issue. Improvements in clinical parameters through this procedure will translate into a greater likelihood of long-term tooth retention and an improvement in the patient's quality of life.

In order to achieve this, the following research question will be addressed: What is the efficacy of LPR-F in conjunction with a complete papilla preservation (EPP) technique for the treatment of infrabony periodontal defects in CESA patients in terms of clinical and radiographic periodontal parameters in comparison with the same technique, but without the use of L-PRF? All patients diagnosed with periodontal disease (loss of interproximal clinical attachment loss in 2 non-adjacent teeth or clinical attachment loss of ≥3mm associated with a probing depth of 3 mm in two or more teeth) will be included, who after re-evaluation 6 weeks after non-surgical periodontal therapy presented residual probing depths equal to or greater than 6 mm associated with interproximal intrabony periodontal defects of at least 2 walls, with a depth ≥ 3 mm and an angulation ≤ 40º determined on a periapical radiograph. Patients with underlying untreated pathologies such as diabetes and hypertension, patients taking medications that interfere with the healing process such as bisphosphonates, diseases that alter bone metabolism such as osteoporosis, and pregnant or breastfeeding women will be excluded. 30 patients (30 defects) will be randomly allocated into an interventional group for the treatment of the infrabony defect. One group will be treated with an EPP technique using L-PRF as the defect filling material and the other group will be treated with the same technique, but with no biomaterial to fill the defect.

The clinical parameters that will be evaluated in each group will be: O'Leary Bacterial Plaque Index (PI), bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL), gingival margin position (GMP), distance from the interproximal contact point to the papilla tip (PP), papilla width (PW), and keratinized gingiva width (KW). These parameters will be measured before the surgical procedure and 6 months after surgery.

The radiographic measurements will be obtained by calibrated operators and will be analyzed in all subjects from a CBCT performed before surgical treatment and 6 months postoperatively. The infrabony component of the defect (INFRA) will be measured, allowing the calculation of the defect filling percentage after surgery (%DF). Additionally, measurements of the mesiodistal width (M-D) and buccal-palatal/lingual width (B-P/L) will be obtained. Researchers will evaluate clinical and radiographic parameters at baseline and 6 months post-surgery. Patients will report their level of pain 24 hours and 7 days after surgery.

The relevance of the present study is based on the need in the field of periodontics to find minimally invasive, effective and low-cost surgical techniques with the least amount of post-surgical complications that will successfully treat infrabony defects of teeth affected by severe periodontitis, a growing public health issue. Improvements in clinical parameters through this procedure will result in a greater likelihood of long-term tooth retention and an improvement in quality of life for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontal disease (loss of interproximal clinical attachment loss in 2 non-adjacent teeth or clinical attachment loss of ≥3mm associated with a PD >3 mm in two or more teeth) will be included.
* After re-evaluation (6 weeks after non-surgical periodontal therapy) presented residual probing depths equal to or greater than 6 mm.
* Residual pocket is associated with interproximal intrabony periodontal defects of at least 2 walls, with a depth ≥ 3 mm and an angulation ≤ 40º determined on a periapical radiograph.

Exclusion Criteria:

* Patients with an underlying decompensated pathology such as diabetes and hypertension.
* Patients taking medications that interfere with the healing process such as bisphosphonates.
* Patients with diseases that alter bone metabolism such as osteoporosis.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Probing depth | From enrollment to the end of treatment 6 months postoperatively
  Distance between the gingival margin and the bottom of the periodontal sulcus or pocket.
Clinical attachment level | From enrollment to the end of treatment 6 months postoperatively
  Distance between the cemento-enamel junction (CEJ) or a stable reference to the bottom of the periodontal pocket.
Bleeding on probing | From enrollment to the end of treatment 6 months postoperatively
  It will be evaluated dichotomously in 6 sites per tooth and will be defined as a percentage by dividing the sites that bleed on probing with the total number of sites examined multiplied by 100.
Distance from contact point to tip of papilla (PP) | From enrollment to the end of treatment 6 months postoperatively
  Distance between the interproximal contact point and the tip of the interproximal papilla
Keratinized Gingiva Width | From enrollment to the end of treatment 6 months postoperatively
  Distance between the tip of the interproximal papilla and the mucogingival line.
Infrabony component of the defect (INFRA) | From enrollment to the end of treatment 6 months postoperatively
  Determined by the subtraction between distance from CEJ to the bottom of the defect (BD) minus the distance from CEJ to the tip of the interproximal crest (IC)
Defect filling percentage after surgery (%DF) | From enrollment to the end of treatment 6 months postoperatively
  Measured by subtraction between distance from CEJ to the bottom of the defect (BD) minus the distance from CEJ to the tip of the interproximal crest (IC), allowing the calculation of percentage defect filling (%DF) after surgery
Mesiodistal width (M-D) of the defect | From enrollment to the end of treatment 6 months postoperatively
  Distance between the mesial and distal wall of the osseous defect
Buccal-palatal/lingual width (B-P/L) of the defect | From enrollment to the end of treatment 6 months postoperatively
  Distance between the bucal and palatal/lingual wall of the osseous defect in mm.

SECONDARY OUTCOMES:
Patient reported outcome: Pain | 24 hours after surgery and one week after surgery
  The intensity of pain (ordinal categorical variable) will be measured after surgical treatment using a visual analogue measurement scale (VAS) that will consist of a measurement 24 hours after surgery by telephone and one week after surgery in the clinical control.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas G Anwandter, DDS, Principal Investigator — Universidad de Los Andes
Locations (1):
- CESA (centro de salud de la clínica odontológica de la Universidad de los Andes), Santiago, San Bernardo, Chile

IPD SHARING:
Plan to Share IPD: Undecided
In order for the results of study to be published in ICMJE journals some information might be shared.